CLINICAL TRIAL: NCT05400434
Title: The Development and Implementation of a Natural Helpers Program to Increase the Recruitment, Retention, and Engagement of Underserved Families in Parent-Child Interaction Therapy (PCIT)
Brief Title: Natural Helpers and PCIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Children's Trust, Miami FL (Other); ConnectFamilias (Unknown)
Responsible Party: Principal Investigator, Jason Jent, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140839
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Child Behavior; Parenting
Keywords: Community Health Workers; Mental Health Disparities
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: The trial was originally designed as a parallel randomized trial. Due to the coronavirus pandemic, the study has been amended to a non-randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Randomized Standard-PCIT group (Experimental): Participants enrolled in the randomized portion of the study and randomized to receive only Standard PCIT for a maximum of 18 weeks.
  Interventions: Behavioral: Standard Parent-Child Interaction Therapy (PCIT)
- Randomized PCIT plus Natural Helper group (Experimental): Participants enrolled in the randomized portion of the study and randomized to receive PCIT plus Natural Helper for a maximum of 18 weeks.
  Interventions: Behavioral: Standard Parent-Child Interaction Therapy (PCIT); Behavioral: Natural Helpers (NH)
- Opt-out Only Standard PCIT group (Experimental): Participants enrolled in the non-randomized portion of the study and opted in to receive only Standard PCIT for a maximum of 18 weeks.
  Interventions: Behavioral: Standard Parent-Child Interaction Therapy (PCIT)
- Opt-in PCIT plus Natural Helper group (Experimental): Participants enrolled in the non-randomized portion of the study and opted in to receive PCIT plus Natural Helper for a maximum of 18 weeks.
  Interventions: Behavioral: Standard Parent-Child Interaction Therapy (PCIT); Behavioral: Natural Helpers (NH)

INTERVENTIONS:
Behavioral: Standard Parent-Child Interaction Therapy (PCIT) — PCIT is an evidence-based behavioral parenting intervention. It is administered as weekly, one-hour sessions with a bilingual PCIT therapist for 18 weeks in one of three PCIT clinics embedded within neighborhood community agencies or virtually.
Behavioral: Natural Helpers (NH) — Natural helpers are lay people to whom others naturally turn for advice, emotional support, and tangible aid. Families received weekly sessions with a natural helpers in their home or virtually for 30-45 minutes for a maximum of 18 weeks. During sessions, natural helpers work with families to (1) explain parenting principles in a culturally and responsive manner; (2) support them in their skill acquisition; and (3) troubleshoot structural barriers to service and other basic life needs.
  Arms: Opt-in PCIT plus Natural Helper group; Randomized PCIT plus Natural Helper group

SUMMARY:
The purpose of the study is to evaluate the effect of a time-limited (i.e., 18 weeks) community health worker (CHW) intervention, referred to as the Parent Child Interaction Therapy (PCIT) plus natural helper (NH) model, on treatment engagement, retention, and child and caregiver outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Families of children 2 years of age to 12 years of age.
2. Children 2 to 7 years of age with a history of child abuse or neglect and/or child behavior problems or children ages 8 years to 12 years of age with history of or risk for abuse and the child does not exhibit clinically significant behavior problems.
3. At the time of enrollment, participants must agree that, within the upcoming six months, they will not move away to a location where they would no longer be able to regularly attend weekly sessions (i.e., moving out of Miami Dade County).

Exclusion Criteria:

1. Families with child younger than 2 years of age or older than 7 years of age with clinically significant behavior problems
2. Adults who are unable to consent and prisoners

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2026-12-27 (Estimated); Study Completion 2026-12-27 (Estimated)

PRIMARY OUTCOMES:
Child externalizing behavior as measured by ECBI Intensity Scale | Up to 26 weeks
  The Eyberg Child Behavior Inventory (ECBI) is a 36-item caregiver report measure of disruptive behaviors in children ages 2-16 . The Intensity Scale assesses the frequency of behavior problems (1=never to 7=always) with total scores ranging from 36 to 252. A raw score of 131 or higher on the Intensity Scale is considered clinically significant child externalizing behavior.
Child externalizing behavior as measured by ECBI Problem Scale | Up to 26 weeks
  The Eyberg Child Behavior Inventory (ECBI) is a 36-item caregiver report measure of disruptive behaviors in children ages 2-16 . The Problem Scale assesses caregiver perceived behavior problems (1 = yes, 0 = no) with total scores ranging from 0 to 36. A raw score of 15 or higher on the Problem Scale is considered clinically significant child externalizing behavior.
Parenting Skills as measured by the Dyadic Parent-Child Interaction Coding System (DPICS-IV) | Up to 26 weeks
  The DPICS-IV is a behavioral observation tool used to code and assess caregiver behaviors and the quality of caregiver and child interactions. PCIT therapists code the three 5-minute DPICS-IV observations: (1) child-led play (CLP), (2) parent-led play (PLP), and (3) clean-up (CU). The number of positive parenting practices (e.g., labeled praises, reflections, and behavior descriptions) and negative parenting practices are tallied (e.g., questions, commands, and criticisms) are coded during CLP observations. During PLP and CU observations, caregiver verbalizations were coded to generate rates of: (1) caregiver effective commands, (2) caregiver correct follow-through on effective commands, and (3) child compliance to effective commands. The higher the score the higher the parenting behavior and child compliance.
Parenting Stress as measured by Parenting Stress Index Short Form (PSI-SF-4) | Up to 26 weeks
  The PSI-SF-4 is a 36-item self-report questionnaire used to measure caregiver stress and difficulties in the caregiver-child relationship for caregivers of youth between ages 0-12. The PSI-SF-4 yields a Total Stress percentile score (0-100) with higher scores indicating higher stress.
Family conflict as measured by Bloom's Family Processes Scale | Up to 26 weeks
  The Bloom's Family Processes Scale assesses family conflict and cohesion using a 5-item conflict subscale (e.g. "we fight a lot in our family"). Caregivers rate their level of agreement on a five-point Likert scale (1=strongly agree to 5=strongly disagree). Total score ranges from 5-25 with the higher scores indicating greater conflict.
Family cohesion as measured by Bloom's Family Processes Scale | Up to 26 weeks
  The Bloom's Family Processes Scale assesses family cohesion using a 5-item cohesion subscale (e.g., "there is a feeling of togetherness in our family"). Caregivers rate their level of agreement on a five-point Likert scale (1=strongly agree to 5=strongly disagree). Total score ranges from 5-25 with the higher scores indicating greater cohesion.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Jent, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - ConnectFamilias, Miami, Florida
  - Mailman Center for Child Development, Miami, Florida

IPD SHARING:
Plan to Share IPD: No